CLINICAL TRIAL: NCT03455283
Title: A Study of Pattern of Use for Gadolinium-Based Contrast Agents (GBCAs) in Patients Undergoing Contrast-Enhanced Magnetic Resonance (CE-MR) Examination - A Prospective, Multicenter, Observational Study
Brief Title: Post-marketing Safety Study in Participants of All Pathologies Who Receive Gadolinium-Based Contrast Agents (GBCAs) for Contrast-Enhanced Magnetic Resonance Imaging (MR) Examination
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CLA-17-01; EUPAS21473 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Magnetic Resonance Imaging (MRI)
MeSH Terms: interventions — ferumoxtran-10

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clariscan 0.5 mmol/ml: Participants will receive Clariscan 0.5 mmol/ml injection as apart of clinical practice at the medical discretion of the prescribing physician.
  Interventions: Drug: Clariscan
- All Gadolinium-Based Contrast Agents (GBCAs): Participants will receive GBCA as part of clinical practice at the medical discretion of the prescribing physician.
  Interventions: Other: Gadolinium-Based Contrast Agents

INTERVENTIONS:
Drug: Clariscan — Clariscan 0.5 mmol/ml solution for injection will be administered as part of clinical practice according to the judgment of the site with regard to medical need.
  Groups: Clariscan 0.5 mmol/ml
Other: Gadolinium-Based Contrast Agents — All GBCAs will be selected by the sites and recorded as by the brand names.
  Groups: All Gadolinium-Based Contrast Agents (GBCAs)

SUMMARY:
The purpose of this study is to prospectively collect data on the pattern of use for gadolinium-based contrast agents (GBCAs) in real-life setting with special reference to Clariscan after its commercial launch in Europe and in addition quality of images, diagnostic confidence and customer satisfaction will be assessed on a Likert scale by the local radiologist/technician and spontaneously reported immediate and delayed adverse events (AEs) to assess the effectiveness and safety profile of GBCAs in clinical practice respectively.

ELIGIBILITY:
Inclusion Criteria: Participants may be included in the study if they meet all of the following criteria:

* Participants of all ages and both male/females
* Participants of all pathologies who require contrast-enhanced magnetic resonance (CE-MR) imaging as part of their diagnostic work up and the radiologist/physician has made the decision to use extracellular gadolinium-based contrast agents (GBCAs) as part of routine clinical practice
* Participants Who Provide informed consent to participate in study

Exclusion Criteria:

* Use of liver-specific GBCAs (Primovist and MultiHance when used for liver excretion properties)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants routinely evaluated with CE-MR in one of 17 European radiology centres. Eligible centres will have Clariscan included on the formulary for Magnetic resonance (MR) examinations and have electronic record of cumulative data and are willing to report the cumulative data at the end of the recruitment period. Only one investigator per centre will be selected to perform the MR examination for that centre as part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 2118 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Pattern of Use of GBCAs in Magnetic Resonance Imaging (MRI) Centres | Up to 3 months
  The Pattern of use will be assessed on summary data collected from: number of radiological procedures (including ultrasound, MR, computed tomography [CT] scan, fluoroscopy, X-ray, single-photon emission CT [SPECT], and positron emission tomography [PET] examinations), number of MR machines, number of enhanced and non-enhanced procedures, characteristics of the treated population (age, gender, BMI), dose indication, referring physician (seniority or specialty) performed by the study centre, investigator and patient-level variables. A qualitative analysis of these variables will be performed describing the overall pattern of use, referral pattern, and challenges in a radiological practice.

SECONDARY OUTCOMES:
Quality of Visualization of the Contrast-Enhanced Magnetic Resonance (CE-MR) Image, Based on the Local Radiologist Assessment | Post-image acquisition on Day 1
  Quality of image will be assessed by the local reporting radiologist on a 4-point Likert scale. For cardiovascular magnetic resonance angiography (MRA), qualitative assessment will be performed by blinded readers and assess image quality on a scale of 1 to 4 as 1=poor image quality and blurring of the arterial segment; 2=fair image quality, inadequate arterial enhancement for confident diagnosis; 3=good image quality and arterial enhancement, adequate for confident diagnosis; 4=excellent image quality and arterial enhancement, for highly confident diagnosis. For Magnetic resonance imaging (MRI), characterisation of the lesion (or most representative lesion, i.e., enhancing and/or largest if there will be >1 lesion present) will be assessed on a 4-point scale as 1= poor, inadequate; 2= fair, partial; 3= good, adequate; 4= excellent.
Change in Diagnostic Confidence (Evaluated by Local Radiologist) in Pre-Contrast and Post-Contrast CE-MR Examination Results | Pre and post administration on Day 1
  For each participant based on the most representative lesion. All available sequences (e.g., fluid attenuation inversion recovery [FLAIR], T2, and T1 with and without contrast administration) will be available for readers to review and evaluate. Before reviewing the CE-MR image, the radiologist will be asked to enter the confidence to make a diagnosis for the participant as a whole number between 0% to 100% based only on the non-enhanced image. The radiologist will then enter the diagnostic confidence as a whole number between 0% to 100% after the CE-MR scan results are read. This will be used to calculate the change in diagnostic confidence in this study by the local radiologist for all GBCAs including Clariscan.
Customer Satisfaction Survey, Based on the Reports by the Local Nurse/Radiology Technician | Upto end of recruitment (upto 90 days)
  Customer satisfaction survey was reported once per centre by MR nurse/technician from the investigator's staff - Quality of packaging including bottles, syringe, marking, pack size available. This will be recorded once for each GBCA used at the study centre as an overall impression and rated as: 1 = can be improved; 2 = good; 3 = excellent.
Percentage of Participants With Treatment-Related Adverse Events (AEs) | Up to 3 months

OTHER OUTCOMES:
Quality of Visualization of the Contrast-Enhanced Magnetic Resonance (CE-MR) Image, Based on the Assessment by MR Experts | Within 18 months from study start date
  The anonymised images will be blindly analysed by an expert MR radiologist panel to assess the quality of images. The first 50 images will be analysed in a 1:1 ratio for Clariscan and other GBCAs, i.e., the first consecutive 25 images for Clariscan and the first consecutive 25 images of the other GBCAs (excluding liver-specific GBCAs). This analysis will be performed at a later date and not part of the initial read out of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Radiology and Nuclear Medicine Ludwigshafen, Otto-Stabel Str. 2-4, Ludwigshafen, Germany
- University of Oslo, Division of Radiology and Nuclear Medicine, P.O. Box 1072, Blindern, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No